CLINICAL TRIAL: NCT04755595
Title: Combination Facial Aesthetic Treatment in Millennials
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Principal Investigator, Jared Jagdeo, MD, MS, Associate Professor of Dermatology, State University of New York - Downstate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1547415
Record Dates: First submitted 2021-01-25; First posted 2021-02-16 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Dermatological Non-Disease
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, rater-blinded, pilot study to evaluate patient satisfaction with facial aesthetic treatment using a combination of botulinum toxin and dermal fillers. The three types of injectables are Botox Cosmetic (onabotulinumtoxinA), Juvéderm Voluma XC (hyaluronic acid gel filler), and Juvéderm Volbella XC (hyaluronic acid gel filler). Twenty individuals who belong to the millennial generation and meet eligibility criteria will be enrolled. Study participants will receive all three injectables during a single procedure. The primary endpoint is the change in satisfaction after facial aesthetic treatment, using the FACE-Q Satisfaction with Facial Appearance Overall Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Facial aesthetic treatment (Experimental): Study participants will receive all three injectables: Botox Cosmetic (onabotulinumtoxinA), Juvéderm Voluma XC (hyaluronic acid gel filler), and Juvéderm Volbella XC (hyaluronic acid gel filler) during a single procedure, with an optional touch-up treatment at 2 weeks.
  Interventions: Drug: Botox Cosmetic Injectable Product; Device: Juvéderm Voluma XC; Device: Juvéderm Volbella XC

INTERVENTIONS:
Drug: Botox Cosmetic Injectable Product — Acetylcholine release inhibitor and a neuromuscular blocking agent
  Other Names: onabotulinumtoxinA
Device: Juvéderm Voluma XC — Gel implants consisting of cross-linked hyaluronic acid
Device: Juvéderm Volbella XC — Gel implants consisting of cross-linked hyaluronic acid

SUMMARY:
With 63% of consumers willing to consider investing in facial aesthetics and 73% of consumers worldwide expecting to invest in aesthetic treatments in the upcoming year, it is imperative to explore patient satisfaction and psychosocial impact of a multimodal aesthetic treatment in a millennial cohort. The investigators hypothesize that a combination approach to facial aesthetic treatment in a millennial cohort will result in increased patient-reported satisfaction in multiple areas, including perception of aging concerns and quality of life.

DETAILED DESCRIPTION:
This is a single-center, prospective, rater-blinded, pilot study to evaluate patient satisfaction with facial aesthetic treatment using a combination of botulinum toxin and dermal fillers. The three types of injectables are Botox Cosmetic (onabotulinumtoxinA), Juvéderm Voluma XC (hyaluronic acid gel filler), and Juvéderm Volbella XC (hyaluronic acid gel filler). Twenty individuals who belong to the millennial generation (i.e., born between January 1, 1981 and December 31, 1996)1 and meet eligibility criteria will be enrolled. Study participants will receive all three injectables during a single procedure, with an optional touch-up treatment at 2 weeks. The primary endpoint is the change in satisfaction after facial aesthetic treatment, using the FACE-Q Satisfaction with Facial Appearance Overall Scale. Other outcome measures include various FACE-Q Aesthetic scales, digital skin imaging analysis, photographs, and rater-blinded clinical assessment using the Global Aesthetic Improvement Scale (GAIS).

ELIGIBILITY:
Inclusion Criteria:

* Date of birth between January 1, 1981 and December 31, 1996
* Naiveté to facial injections of botulinum toxin and dermal filler
* Desire to receive all three facial cosmetic injectables in the study
* Suitable candidate to receive facial injectables, as determined by clinician judgment
* Provision of written informed consent for all study procedures
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Desire to receive only one or two of the facial injectables
* Dermatologic or medical conditions at the injection sites that may be exacerbated by the study procedures (e.g., severe acne, active infection, open sores or lesions, history of cold sores)
* Pre-existing cardiovascular disease (e.g., heart failure, coronary artery disease)
* Pre-existing swallowing or respiratory disorders (e.g., dysphagia, asthma, COPD)
* Peripheral motor neuropathy disease, amyotrophic lateral sclerosis, or neuromuscular junctional disorders (e.g., myasthenia gravis, Lambert-Eaton syndrome)
* Known hypersensitivity or allergies to any of the components of the administered drugs/devices in the study (e.g., Gram-positive bacterial proteins, lidocaine)
* History of anaphylaxis or multiple severe allergies
* History of a bleeding or coagulation disorder
* Pregnant or breast-feeding
* Current and/or scheduled use of the following medications: immunosuppressants, anticoagulants (e.g., warfarin, heparin, rivaroxaban), antiplatelets (e.g., clopidogrel, ticagrelor, NSAIDs), antibiotics (e.g., aminoglycosides), anticholinergics, muscle relaxants
* Procedures or treatments to the face in the past 14 days (e.g., chemical peel, laser surgery, microdermabrasion)
* Plan to undergo elective cosmetic procedure on the face (e.g., laser surgery, plastic surgery, physician-strength chemical peel) during the study
* Any medical condition(s) that could be compromised by participating in the study

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD, MS, Principal Investigator — SUNY Downstate Medical School
Locations (1):
- SUNY Downstate Health Sciences University, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Facial Aesthetic Treatment
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Facial Aesthetic Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 13
  White, Hispanic | 2
  Asian | 3
  Two or more races | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: FACE-Q Satisfaction With Facial Appearance Overall Scale
Description: To assess changes in patient's satisfaction with their appearance following a combination facial aesthetic treatment, using the FACE-Q Satisfaction with Facial Appearance Overall Scale. This tool consists of several questions. For each question, the study participant selects a number from 1 to 4. Higher number are associated with higher satisfaction with facial appearance. The raw scores of the primary outcome measure were transformed by the Rasch measurement method into a 0-to-100 point scale.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of satisfaction of overall facial appearance.
- Post-treatment: Post-treatment assessment of satisfaction of overall facial appearance (conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 42.35 (8.94) | 59.42 (15.08)

2. Secondary Outcome: FACE-Q Appraisal of Lines Overall
Description: To assess changes in patient dissatisfaction with the appearance of overall facial lines, using the FACE-Q Appraisal of Lines: Overall Scale. The tool consists of ten questions regarding self-perception of overall facial lines. For each question, study participants select a number from 1 to 4, with higher numbers reflecting greater dissatisfaction with facial lines. The total score is tallied. The minimum total score is 10 and the maximum total score is 40. A higher total score is associated with greater dissatisfaction with facial lines. The mean total score at baseline and 2 months post procedure are reported.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of dissatisfaction with facial lines.
- Post-treatment: Post-treatment assessment of dissatisfaction with facial lines (conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 21.5 (6.8) | 15.1 (3.2)

3. Secondary Outcome: FACE-Q Expectations Scale
Description: To assess patient expectations regarding the impact of facial aesthetic treatment on their lives, using the FACE-Q Expectations Scale. This tool consists of eight statements. For each statement, the study participant selects a number from 1 to 4, where 1 represents "definitely disagree", 2 represents "somewhat disagree", 3 represents "somewhat agree", and 4 represents "definitely agree". The total score of the statements is tallied. The minimum total score is 8 and the maximum total score is 32. The higher the total score, the greater positive impact the participants believe the treatments will have on their lives. The mean total score at baseline is reported.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Assessment of expectations regarding the impact of facial aesthetic treatment on participants' lives
Arm/Group | Baseline
Number analyzed (Participants) | 20
score on a scale | 17.4 (4.6)

4. Secondary Outcome: FACE-Q Social Function Scale
Description: To assess changes in psychosocial factors after facial aesthetic treatment, using FACE-Q Social Function Scale. This tool consists of eight statements. For each statement, the study participant selects a number from 1 to 4, where 1 represents "definitely disagree", 2 represents "somewhat disagree", 3 represents "somewhat agree", and 4 represents "definitely agree". The total score of the statements is tallied for each patient. The minimum total score is 8 and the maximum total score is 32. A higher total score reflects greater social functioning. The mean total score is reported at baseline and 2 months after the procedure.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of social function
- Post-treatment: Post-treatment assessment of social function (conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 24.4 (4.6) | 27.4 (4.3)

5. Secondary Outcome: FACE-Q Patient-Perceived Age Visual Analogue Scale
Description: To assess changes in self-perceived age after facial aesthetic treatment, using the FACE-Q Patient-Perceived Age Visual Analogue Scale. The study participant selects a number on the scale from -15 to +15. 0 corresponds to "I look my age". -15 corresponds to "I look 15 years younger". +15 corresponds to "I look 15 years older". The mean score at baseline and 2 months post procedure are reported.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of self-perceived age
- Post-treatment: Post-treatment assessment of self-perceived age (conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 0.2 (2.3) | -2.2 (3.1)

6. Secondary Outcome: FACE-Q Satisfaction With Cheeks
Description: To assess changes in patient satisfaction with the appearance of their cheeks after facial aesthetic treatment, using the FACE-Q Satisfaction with Cheeks Scale. The tool consists of five questions regarding self-perception of cheeks. For each question, study participants select a number from 1 to 4, with higher numbers reflecting greater satisfaction with cheeks. The total score is tallied. The minimum total score is 5 and the maximum total score is 20. A higher total score is associated with greater satisfaction with cheeks. The mean total score at baseline and 2 months post procedure are reported.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of satisfaction of cheeks.
- Post-treatment: Post-treatment assessment of satisfaction of cheeks (conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 13.3 (3.4) | 16.9 (2.1)

7. Secondary Outcome: FACE-Q Satisfaction With Outcome Scale
Description: To assess patient satisfaction with facial aesthetic treatment, using the FACE-Q Satisfaction with Outcome Scale. This tool consists of six statements. For each statement, the study participant selects a number from 1 to 4, where 1 represents "definitely disagree", 2 represents "somewhat disagree", 3 represents "somewhat agree", and 4 represents "definitely agree". The total score is tallied. The minimum total score is 6 and the maximum total score is 24. A higher total score is associated with greater satisfaction with outcome. The mean total score 2 months after the procedure is reported.
Time Frame: 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Post-treatment: Post-treatment assessment of satisfaction with outcome(conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Post-treatment
Number analyzed (Participants) | 19
score on a scale | 20.8 (2.9)

8. Secondary Outcome: FACE-Q Psychological Function Scale
Description: To assess changes in psychosocial factors after facial aesthetic treatment, using the FACE-Q Psychological Function Scale. This tool consists of ten statements. For each statement, the study participant selects a number from 1 to 4, where 1 represents "definitely disagree", 2 represents "somewhat disagree", 3 represents "somewhat agree", and 4 represents "definitely agree". The total score is tallied. The minimum total score is 10 and the maximum total score is 40. A higher total score is associated with better psychological functioning. The mean total score at baseline and 2 months after the procedure are reported.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of psychological function
- Post-treatment: Post-treatment assessment of psychological function(conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 30.5 (8.2) | 34.9 (5.1)

9. Secondary Outcome: FACE-Q Aging Appraisal Scale
Description: To assess changes in self-perceived age after facial aesthetic treatment, using the FACE-Q Aging Appraisal Scale. This tool consists of seven statements. For each statement, the study participant selects a number from 1 to 4, where 1 represents "definitely disagree", 2 represents "somewhat disagree", 3 represents "somewhat agree", and 4 represents "definitely agree". The total score is tallied. The minimum total score is 7 and the maximum total score is 28. A lower total score is associated with greater satisfaction with self-perceived age. The mean total score at baseline and 2 months after the procedure are reported.
Time Frame: 2 months after the procedure compared to baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 12.6 (5.6) | 9.8 (4.8)

10. Secondary Outcome: FACE-Q Satisfaction With Lips
Description: To assess changes in patient satisfaction with the appearance of their lips after facial aesthetic treatment, using the FACE-Q Satisfaction with Lips Scale. The tool consists of ten questions regarding self-perception of lips. For each question, study participants select a number from 1 to 4, with higher numbers reflecting greater satisfaction with lips. The total score is tallied. The minimum total score is 10 and the maximum total score is 40. A higher total score is associated with greater satisfaction with lips. The mean total score at baseline and 2 months post procedure are reported.
Time Frame: Baseline and 2 months after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline assessment of satisfaction with lips.
- Post-treatment: Post-treatment assessment of satisfaction with lips (conducted 2 months post-combination facial aesthetic treatment using soft tissue fillers and botulinum toxin).
Arm/Group | Baseline | Post-treatment
Number analyzed (Participants) | 20 | 19
score on a scale | 25.4 (7.3) | 34.9 (4.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over two months.
Arm/Group | Facial Aesthetic Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Facial Aesthetic Treatment (N=20)
Bruising (Skin and subcutaneous tissue disorders) | 9
Edema (Skin and subcutaneous tissue disorders) | 14
Headache (General disorders) | 4
Soreness (General disorders) | 4
Lumps localized to midface dermal filler injection sites (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT04755595/Prot_SAP_000.pdf